CLINICAL TRIAL: NCT03201094
Title: Impact of Neuromuscular Stimulation and High Protein Nutritional Supplementation on Long-term Recovery After Aneurysmal Subarachnoid Hemorrhage.
Brief Title: Impact of NMES and HPRO on Recovery After SAH- Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Neeraj Badjatia, Professor of Neurology, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HP-00074174
Record Dates: First submitted 2017-06-23; First posted 2017-06-28 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Subarachnoid Hemorrhage; Muscle Atrophy; Inflammation; Nutritional and Metabolic Disease
MeSH Terms: conditions — Subarachnoid Hemorrhage; Muscular Atrophy; Inflammation; Metabolic Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Standard of Care (No Intervention): Patients will receive standard of care mobilization and nutritional supplementation throughout the study period.
- HPRO + NMES (Experimental): Patients will receive high protein supplementation(HPRO) administered within 30 minutes after each NMES session and additionally once at approximately 10 PM.
  Interventions: Device: Neuromuscular Electrical Stimulation (NMES); Dietary Supplement: High Protein Supplementation
- NMES only (Experimental): Patients will undergo two 30 minute NMES sessions per day during study period.
  Interventions: Device: Neuromuscular Electrical Stimulation (NMES)
- HPRO only (Experimental): Patients will receive HPRO three times daily during study period
  Interventions: Dietary Supplement: High Protein Supplementation

INTERVENTIONS:
Device: Neuromuscular Electrical Stimulation (NMES) — Neuromuscular electrical stimulation twice daily during study period.
  Arms: HPRO + NMES; NMES only
Dietary Supplement: High Protein Supplementation — High protein supplementation with whey protein shakes taken three times a day during study period.
  Arms: HPRO + NMES; HPRO only

SUMMARY:
The study purpose is to investigate the hypothesis that in adults with SAH, early neuromuscular electrical stimulation (NMES) and high protein supplementation (HPRO) will improve muscle mass, metabolic and inflammatory biomarker profiles, compared to SAH controls receiving standard of care interventions for nutrition and mobilization. The investigators will accomplish this by studying the effects of a high protein (HPRO) nutritional treatment as well as NMES intervention have upon muscle wasting and motor strength acutely after SAH. This will be addressed in a prospective trial of SAH patients receiving HRPO with NMES as compared to age and severity-matched SAH patients undergoing standard of care interventions for nutrition and mobilization. Additionally, the study will investigate the impact HPRO and NMES interventions have upon inflammatory cytokines and markers of energy balance. Results of this study will establish evidence for precision nutrition plus early exercise to mitigate the catabolic and inflammatory state produced by SAH to improve muscle, metabolic, and health recovery outcomes.

ELIGIBILITY:
Inclusion criteria:

1. . Being diagnosed with aneurysmal SAH
2. . Aneurysmal repair within 48 hours of ictus.
3. . Age between 25 and 80 years old. (>=25 years old and <=80 years old)
4. . Expected stay in the NCCU > 72 hours.
5. . Admission Hunt Hess Grade >=2.
6. modified Fisher score >1.

Exclusion criteria:

1. . Subjects diagnosed with SAH from trauma, rupture of an arteriovenous malformation, neoplasm, vasculitis, or other secondary causes;
2. . Unlikely to survive one week post hemorrhage either due to impending brain death or likely request for withdrawal of care;
3. . Unlikely to remain in the ICU for more than 7 days;
4. . Body mass index < 15 or >40 kg/m2;
5. . Allergy to whey protein;
6. . Evidence of lower extremity paresis or spasticity within 48 hours of injury
7. . Pre-morbid modified Rankin Score >1.
8. . Known pregnancy
9. . Presence of active malignancy
10. . Diagnosis of an inflammatory disorder
11. . Presence of a neuromuscular disorder
12. . Diagnosis of chronic renal insufficiency or acute kidney injury (GFR < 30 mL/min/1.73m2)
13. . Hepatic insufficiency defined as AST/ALT levels >2.5 above normal upper limits.
14. . On-going seizure activity as assessed clinically or by electrographic detection on continuous electroencephalogram (cEEG) at time of enrollment
15. . Prisoner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in muscle layer thickness of the quadriceps muscle as measured by muscle ultrasound scan at the end of study period. | 14 days
  Change in the muscle layer thickness of the quadriceps muscle as measured by ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj Badjatia, MD MSc, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No